CLINICAL TRIAL: NCT01569490
Title: Striving to Quit: First Breath Tobacco Cessation Research
Brief Title: Striving to Quit: First Breath
Acronym: STQ FB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-0136
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Smoking Cessation; Smoking; Nicotine Dependence
MeSH Terms: conditions — Smoking Cessation; Smoking; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment incentives (Experimental): Incentives for biochemical verification visits, treatment engagement, and abstinence
  Interventions: Behavioral: Incentives for abstinence and treatment engagement
- Attendance incentive (Active Comparator): Incentives for only attending the biochemical verification visits
  Interventions: Behavioral: Attendance incentive

INTERVENTIONS:
Behavioral: Incentives for abstinence and treatment engagement — Treatment Incentives - incentives for biochemical verification visits, treatment engagement, and abstinence
  Arms: Treatment incentives
Behavioral: Attendance incentive — Attendance Incentives - incentives for only attending the biochemical verification visits
  Arms: Attendance incentive

SUMMARY:
This study is designed to test the hypotheses that incentives can increase both participation in smoking cessation treatment and resulting cessation rates, when they are offered to Medicaid BadgerCare Plus pregnant smokers.

DETAILED DESCRIPTION:
Aim 1: To determine the extent to which contingent financial "treatment incentives" (i.e., incentives for biochemical verification visits, treatment engagement, and abstinence) versus "attendance incentives" (i.e., incentives for only attending the biochemical verification visits), increase rates of prenatal and postnatal smoking abstinence. Participants will be BadgerCare Plus members who are recruited into the First Breath program while pregnant.

Aim 2: To determine the extent to which treatment incentives, versus attendance incentives, increase rates of engagement in First Breath smoking cessation intervention when offered to pregnant and postpartum BadgerCare Plus members.

Aim 3: To determine the cost-effectiveness and reach of the First Breath intervention delivered to pregnant and postpartum smokers when it is paired with treatment incentives and when paired with only attendance incentives.

Aim 4: To determine if the First Breath intervention with treatment incentives, in comparison to that intervention with only attendance incentives, produces significantly greater benefits in pregnant and postpartum women with regards to nonsmoking health outcomes: i.e., reduced depression, increased levels of breast feeding, and greater perceived support.

Aim 5: To identify moderating and mediating effects of treatment incentives when offered in the context of the First Breath intervention delivered to pregnant and postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* enrollment in Wisconsin Medicaid (BadgerCare Plus or Medicaid SSI)
* resides in study area
* member of participating Medicaid HMOs
* not involved in any other stop smoking research studies
* 18 or older
* English speaking
* smoked daily (at least one cigarette each day for at least one week) at some time within the last 6 months
* willingness to quit smoking, cut down, or stay quit
* willing to complete study visits and phone calls
* willing to provide updates in contact information

Exclusion Criteria:

* not enrolled in Wisconsin Medicaid (BadgerCare Plus or Medicaid SSI)
* not enrolled in study area
* not a member of participating Medicaid HMOs
* not pregnant or enrolled in First Breath
* less than 18 years of age
* non-English speaking
* does not smoke daily (at least one cigarette each day for at least one week) at least some time within the last 6 months
* not willing to complete study procedures and assessments or provide updated contact information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3100 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Abstinence from smoking | Measured 6 months after births at follow-up assessment
  The data will be the biochemically confirmed reports of abstinence for the past 7 days (i.e., 7-day point-prevalence abstinence)

SECONDARY OUTCOMES:
Engagement in treatment | Measured 12 months after birth at follow-up assessment
  The primary analyses will compare number of calls and visits completed.
Cost-effectiveness | Measured 12 months after birth
  The primary analysis will contrast the incremental costs of the treatment vs. attendance conditions by computing the Incremental Cost-Effectiveness Ratio (ICER) with regard to attaining 6-month abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B. Baker, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Wisconsin Women's Health Foundation, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Baker TB, Fraser DL, Kobinsky K, Adsit R, Smith SS, Khalil L, Alaniz KM, Sullivan TE, Johnson ML, Fiore MC. A randomized controlled trial of financial incentives to low income pregnant women to engage in smoking cessation treatment: Effects on post-birth abstinence. J Consult Clin Psychol. 2018 May;86(5):464-473. doi: 10.1037/ccp0000278. Epub 2018 Feb 1. PMID 29389142